CLINICAL TRIAL: NCT01489007
Title: Evaluation of Iron Absorption in Healthy Vegetarian Children 4 to 10 Years of Age
Brief Title: Iron Absorption in Vegetarian Children
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Steve Abrams, MD, Professor of Pediatrics, Baylor College of Medicine
Other Study IDs: H-29640
Record Dates: First submitted 2011-12-07; First posted 2011-12-09 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Iron Absorption
Keywords: vegetarian; children; iron; iron absorption

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vegetarian Children: Self-described lacto-ovo vegetarians for the past 6 months (Subjects who include a small amount of fish or chicken in the diet (not more than 2 servings total/week of both combined) will be allowed to participate in this study as these are not major iron contributors to the diet. Subjects must not have eaten any "red meat" however for 6 months.) Control subjects will be non-vegetarians.

SUMMARY:
Few areas are more controversial in pediatric nutrition than the role of a vegetarian diet for children. Advocates make strong health claims whereas others have expressed safety concerns, especially regarding iron nutrition. The frequency of vegetarianism among children is said to be rapidly increasing although clear data are not available. Surveys of children in the US age 8 to 18 reported in the media find that about 3-5% of children are lacto-ovo vegetarian, with some fish or chicken products in the diet. This is a substantial proportion that is very likely to increase over the next few years with essentially no nutrient metabolism data related to this population.

One of the principal concerns with a lacto-ovo vegetarian diet, as preferred by many children, is the lack of heme iron in the diet. A key question that can be evaluated in children is whether iron status is in fact affected by a lacto-ovo vegetarian diet.

According to the American Academy of Pediatrics (AAP Pediatric Nutrition Handbook, 6th Edition, 2008), vegetarian diets can provide appropriate nutrition for children. Depending on the level of dietary restriction, fortified foods or supplements may be necessary during different life stages. In addition, strict vegetarian children may have slightly higher protein needs compared to non-vegetarian children due to decreased protein digestibility in certain plants. The AAP further recommends that children 4-8 years old consume a minimum of five servings per day of beans/nuts/seeds/eggs and six servings per day of calcium-rich foods.

To evaluate this issue, the investigators will use a stable isotope method to directly assess iron status. It is increasingly recognized that the ability to absorb iron when given with vitamin C is a highly accurate measurement of iron status and may be a true gold standard in this regard. In this planned study, investigators will be able to assess both reference dose iron absorption and standard biochemical markers of iron status in a group of lacto-ovo vegetarians and compare them with age- and gender-matched children on a non-vegetarian diet. These data can be important in determining if iron status is decreased in lacto-ovo vegetarians and will serve as a basis for future interventions and evaluations if a difference is found.

DETAILED DESCRIPTION:
Iron absorption studies will be done in 30 healthy vegetarian children 4 to 10 yrs of age and 30 healthy non-vegetarian children who are age and gender matched controls (from another study).

Visit 1: At the time of enrollment, subjects and their families will be asked to come to the General Clinical Research Center (GCRC) of Texas Children's Hospital or the Metabolic Research Unit (MRU) at the Children's Nutrition Research Center for a screening visit. Prior to this visit, demographics from the parent/guardian will be recorded including the child's approximate height and weight, and the study dietitian will obtain two 24-hour dietary recalls from the parent to determine dietary intake for enrollment. During this screening visit, informed written consent will be obtained and anthropometry and vital signs will be recorded.

The study dietitian will instruct the parent/guardian and child on the use of a food scale to weigh and record dietary intake for a 3-day period (ie, 3-day weighed diet record). The 3-day weighed diet record will begin the following day. Upon analysis of their child's intake, parents will be instructed to maintain a similar nutrient intake throughout the study. Compliance will be monitored via 3-day weighed home diet records timed with their other study visits. If analysis shows that the child's intake has significantly changed (± 20% of a nutrient), the parent will be counseled by the study dietitian on readjusting the child's intake back to the usual level determined at baseline.

Visit 2: Subjects will be admitted to the GCRC or MRU as an outpatient after a 2-3h fast and given a reference dose of 1mg iron-58 sulfate as an aqueous solution with 50mg ascorbic acid. They will be observed for 2h after this dose and water will be freely available. No food will be allowed however water is allowed. After 2h subjects will be discharged home and food allowed. After discharge, subjects will record dietary intake using another 3-day weighed diet record.

Visit 3: Prior to this visit, subjects will receive a food scale and will perform another 3-day weighed diet record to demonstrate consistency of diet throughout the study period. Two weeks (+/- 3 days) later subjects will be readmitted and 10mL blood (2 tsp) will be drawn for measurement of iron nutritional parameters (e.g. hepcidin, ferritin, iron, TIBC, transferrin saturation, hemoglobin, hematocrit, and RBC indices) and iron isotope ratio measurement. Labs for iron nutritional parameters may be sent to the TCH Lab or an outside commercial lab. Incorporation of iron-58 will be used to measure absorption from the reference dose (a measure of iron status). Topical numbing cream or spray to minimize pain at the injection site will be offered to all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Delivery at > or = 35.0 weeks gestation with birth weight > or = 2.5 kg
* BMI: 10th - 90th percentile for age and gender
* Ages 4.0 to 10.9 years
* Ethnic distribution of greater Houston area
* Self-described lacto-ovo vegetarians for the past 6 months (Subjects who include a small amount of fish or chicken in the diet (not more than 2 servings total/week of both combined) will be allowed to participate in this study as these are not major iron contributors to the diet. Subjects must not have eaten any "red meat" however for 6 months.) Control subjects will be non-vegetarians.
* Any regularly taken (daily) iron supplements (with or without vitamin D) must be stopped at least 1 month before starting the study. Supplements of vitamin D with calcium, B12, and folate are allowed.

Exclusion Criteria:

* History of any chronic illness.
* Regularly taken (daily) medications (except seasonal allergies).
* Avoidance of dairy products in the diet (controls excluded).
* Females: has had first menstrual period.
* Control subjects will be non-vegetarians whose usual diet includes 2 servings/week or more of red meat.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Effect of vegetarian diet on iron status | At the final study visit (approximately 3-4 weeks after the start of the study)
  At the final study visit, 10 mL blood (2 tsp) will be drawn for measurement of iron nutritional parameters (e.g. hepcidin, ferritin, iron, TIBC, transferrin saturation, hemoglobin, hematocrit, and RBC indices) and iron isotope ratio measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Abrams, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine / Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Thane CW, Bates CJ, Prentice A. Risk factors for low iron intake and poor iron status in a national sample of British young people aged 4-18 years. Public Health Nutr. 2003 Aug;6(5):485-96. doi: 10.1079/PHN2002455. PMID 12943565
- [Background] Craig WJ, Mangels AR; American Dietetic Association. Position of the American Dietetic Association: vegetarian diets. J Am Diet Assoc. 2009 Jul;109(7):1266-82. doi: 10.1016/j.jada.2009.05.027. PMID 19562864